CLINICAL TRIAL: NCT05425823
Title: Randomized Controlled Trial Of A Health Belief Model-Based Intervention To Prompt To Take Up The Childhood Vaccines And Effect On Vaccination Attitudes
Brief Title: Intervention to Promote Childhood Vaccinations and Influence Vaccination Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Kübra Sultan Dengiz, Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 221430001
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Vaccine Hesitancy; Childhood Vaccination
Keywords: Vaccine hesitancy; childhood vaccination; health belief model; parental attitudes; education
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: parallel randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Education and message (Experimental): In Intervention Group 1, a face-to-face training session based on the Health Belief Model will be given once a week and SMS-based short messages will be sent to the spouse.
  Vaccination rates of children in the intervention group-1 in the study at the end of the 1st, 6th and 12th months will be evaluated. Public Attitudes Towards Vaccination Scale-Health Belief Model sub-dimensions (severity, susceptibility, benefit, barrier, health motivation) scores of the intervention group-1 at the 1st, 6th, and 12th months after birth will be evaluated.
  Interventions: Other: Health Belief Model Based Intervention
- Education (Experimental): In Intervention Group 2, face-to-face training will be provided one day a week based on the Health Belief Model.
  Vaccination rates of children in the intervention group-2 in the study at the end of the 1st, 6th and 12th months will be evaluated. Public Attitudes Towards Vaccination Scale-Health Belief Model sub-dimensions (severity, susceptibility, benefit, barrier, health motivation) scores of the intervention group-2 at the 1st, 6th, and 12th months after birth will be evaluated.
  Interventions: Other: Health Belief Model Based Intervention
- Standard Care Group (No Intervention): Standard information about childhood vaccines will be provided to the Standard Care Group at the Family Health Care Center.
  Vaccination rates of children in the Standard Care Group in the study at the end of the 1st, 6th and 12th months will be evaluated. Public Attitudes Towards Vaccination Scale-Health Belief Model sub-dimensions (severity, susceptibility, benefit, barrier, health motivation) scores of the Standard Care Group at the 1st, 6th, and 12th months after birth will be evaluated.

INTERVENTIONS:
Other: Health Belief Model Based Intervention — In intervention group-1, Information Form and PAVS-HBM will be applied as a pre-test to pregnant women who have completed their 28th gestational week. Childhood Vaccination Training Based on the Health Belief Model will be given in the prenatal period by organizing 2 face-to-face and individual sessions for the researcher's pregnant women. Each session will take approximately 30-45 minutes, with each session being in a different week. In addition, at the end of each session, HBM-based short messages will be sent to the pregnant woman's husband and recorded with the Short Message Tracking Form. Intervention group-2 will receive the same training, but no text messages will be sent.
  Arms: Education; Education and message

SUMMARY:
This study aims to determine the effect of pregnant women aged 18 years and older who have completed their 28th week of pregnancy and received intervention based on the Health Belief Model, on encouraging childhood vaccinations and influencing their vaccination attitudes, compared to pregnant women who receive standard care group. The 12-month vaccination rate of newborns and the change in their attitudes will be determined according to the Public Attitude Towards Vaccination Scale - Health Belief Model.

DETAILED DESCRIPTION:
Today, vaccines are still recognized as one of the most important public health services, and millions of lives are saved each year. Despite the success of vaccination, such as eradicating certain diseases in the community and preventing epidemics, it is the fact that approximately 20 million infants/children have insufficient access to vaccines every year. The main reasons for this are vaccine hesitancy or vaccine rejection. Deaths from measles decreased by 73% worldwide between 2000 and 2018, preventing an estimated 23.2 million deaths. According to the Extended Immunization Program in our country, 13 routine vaccines in total are provided free of charge by primary health care services. According to the results of the Turkey Demographic and Health Surveys, the minimum vaccinations required for 12-23 month old children to be deemed to have received all age-appropriate vaccines are as follows; one dose of tuberculosis vaccine, three doses of pertussis-tetanus-polio-hemophilus influenza type b vaccine, three doses of hepatitis b vaccine, three doses of pneumococcal conjugate vaccine, one dose of oral polio vaccine. Considering both the vaccination card of the children (59%) and the personal statements (8%) of the mothers in our society, it was determined that only 67% of the children aged 12-23 months received all age-appropriate vaccinations. In addition, 2% of 12-23-month-old children have never been vaccinated. In addition, 50% of 24-35 months old children have all their age-appropriate vaccinations, while 3% have never been vaccinated. Looking at all these rates, it is seen that some babies/children are not vaccinated for various reasons, even in our country alone. To increase vaccination rates, preventive interventions should be developed to identify the causes of vaccine hesitations and reduce these hesitations. What needs to be done first to eliminate vaccine hesitations should be to increase the perceived sensitivity of individuals to the vaccine and decrease their expectations for negative results. At the same time, it is necessary to know the factors that cause negative attitudes about vaccination and to make them positive so that attitudes can turn into behaviors. According to the Health Belief Model, which is one of the models related to the development and maintenance of health behaviors, the probability of a person taking action to prevent the disease depends on the perceived susceptibility, perceived severity, perceived benefit, and perceived barrier factors, and indirectly includes the probability of exhibiting preventive health behavior. Among the factors affecting the vaccination decision of pregnant women, vaccine risk perceptions are effective; It has been determined that pregnant women who have general knowledge about the vaccine, those who know that there is a national vaccination policy, and those who believe that the vaccine is beneficial for their babies are more likely to be vaccinated. For this reason, it is recommended that the advice of healthcare professionals should be personalized. In line with all these data, the aim of the study is to examine the effectiveness of the intervention of training to be given to pregnant women about childhood vaccinations and sending messages to their spouses within the framework of the Health Belief Model; to evaluate the effect on childhood vaccination rates and vaccination attitudes in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* The pregnant woman and her spouse are Turkish literate,
* Completing the 28th week of pregnancy,
* Desire to participate in the study,
* The pregnant's spouse has any type of mobile phone.

Exclusion Criteria:

* The pregnant woman has any mental problem that causes learning difficulties or has been diagnosed (if detected in the pregnancy outpatient clinic record).
* 38 weeks of pregnancy and above
* Living outside of the 3 central districts of Konya (Selçuklu, Meram, Karatay)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy, completing the 28th week of pregnancy
Enrollment: 54 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Children's vaccination rates 1st | 1.month
  Childhood vaccination rates of intervention groups and standard care group in the study were similar at the end of the 1st month.
Children's vaccination rates 6th | 6th.month
  Childhood vaccination rates of intervention groups and standard care group in the study were similar at the end of the 6th month.
Children's vaccination rates 12th | 12.month
  Childhood vaccination rates of intervention groups and standard care group in the study were similar at the end of the 12th months.

SECONDARY OUTCOMES:
Scores from the Public Attitude Towards Vaccination Scale - Health Belief Model | 1.month
  The Public Attitude Towards Vaccination Scale-Health Belief Model sub-dimensions (severity, susceptibility, benefit, barrier, health motivation) scores of the intervention groups (1 and 2) were similar the standard care group's at the 1st months postpartum.
  Evaluation of the scale cannot be made over the total score. It consists of a total of 26 questions and 5 sub-dimensions. When all five sub-dimensions and sub-dimensions with a five-point Likert response are evaluated separately; Susceptibility and severity sub-dimension consists of 4 items (lowest 4, highest 20 points), benefit and health responsibility sub-dimension 5 items (lowest 5 points, highest 25 points), barrier sub-dimension consists of 8 items (lowest 8, highest 40 points). While a decrease in the score in the obstacle sub-dimension indicates a positive attitude, an increase in the score in the other sub-dimensions indicates a positive attitude.
Scores from the Public Attitude Towards Vaccination Scale - Health Belief Model | 6.month
  The Public Attitude Towards Vaccination Scale-Health Belief Model sub-dimensions (severity, susceptibility, benefit, barrier, health motivation) scores of the intervention groups (1 and 2) were similar the standard care group's at the 6th months postpartum.
  Evaluation of the scale cannot be made over the total score. It consists of a total of 26 questions and 5 sub-dimensions. When all five sub-dimensions and sub-dimensions with a five-point Likert response are evaluated separately; Susceptibility and severity sub-dimension consists of 4 items (lowest 4, highest 20 points), benefit and health responsibility sub-dimension 5 items (lowest 5 points, highest 25 points), barrier sub-dimension consists of 8 items (lowest 8, highest 40 points). While a decrease in the score in the obstacle sub-dimension indicates a positive attitude, an increase in the score in the other sub-dimensions indicates a positive attitude.
Scores from the Public Attitude Towards Vaccination Scale - Health Belief Model | 12.month
  The Public Attitude Towards Vaccination Scale-Health Belief Model sub-dimensions (severity, susceptibility, benefit, barrier, health motivation) scores of the intervention groups (1 and 2) were similar the standard care group's at the 12th months postpartum.
  Evaluation of the scale cannot be made over the total score. It consists of a total of 26 questions and 5 sub-dimensions. When all five sub-dimensions and sub-dimensions with a five-point Likert response are evaluated separately; Susceptibility and severity sub-dimension consists of 4 items (lowest 4, highest 20 points), benefit and health responsibility sub-dimension 5 items (lowest 5 points, highest 25 points), barrier sub-dimension consists of 8 items (lowest 8, highest 40 points). While a decrease in the score in the obstacle sub-dimension indicates a positive attitude, an increase in the score in the other sub-dimensions indicates a positive attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz S Hisar, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Konya/MEram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No